CLINICAL TRIAL: NCT06721234
Title: Role of Femoral Vein Wall Thickness and Inflammatory Markers in Patients With Behcet Disease
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Engy Louis Fawzy, Principal investigator, Sohag University
Other Study IDs: Soh-Med--24-11-03MS
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-11

CONDITIONS: Behçet
MeSH Terms: conditions — Behcet Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluation of femoral vein wall thickness and inflammatory indices in patients with Behcet disease and assessment of their relation to the disease activity and related some clinical manifestations

ELIGIBILITY:
Inclusion Criteria:

* Patients fulfill the International Criteria for Behcet's Disease (ICBD)
* Age above 18 years old
* Patients cooperative and can answer questions
* Patients who are able and willing to give informed consent

Exclusion Criteria:

* Other rheumatological and vascular diseases
* Patients with abnormal hepatic or renal function tests , hyperlipidemia and impaired coagulation tests
* Patients with hypertension , diabetes mellitus , malignant and active infectious diseases
* Patients who are using aspirin and other platelet active drygs during the previous 6 months
* patients who are not able and willing to give written consent

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12-02 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Femoral Vein Wall thickness | One week

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university, Sohag, Egypt